CLINICAL TRIAL: NCT07075055
Title: Impact of a New Bioceramic Based Intracanal Medication on Postoperative Pain and Periapical Healing
Brief Title: Impact of a New Bioceramic Based Intracanal Medication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hanaa Ewas Korany Mabrouk, Assistant lecturer of Endodontics at Nahda University,, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intracanal Bioceramic
Record Dates: First submitted 2025-07-02; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metapaste Calcium Hydroxide (Active Comparator): About 13 healthy patients of both genders presented with periapical radiolucency will subject to complete preparation of the root canal system using the (Metapaste Calcium Hydroxide(Pre-mixed paste) as an intracanal medicament.
  Interventions: Other: Metapaste Calcium Hydroxide
- Bio C-Temp (Active Comparator): About 13 healthy patients of both genders presented with periapical radiolucency will subject to complete preparation of the root canal system using the (Bio C-Temp) as an intracanal medicament.
  Interventions: Other: Bio C-Temp

INTERVENTIONS:
Other: Metapaste Calcium Hydroxide — To compare the effect of calcium hydroxide and Bio-C Temp as intra canal medications on postoperative pain via VAS and periapical healing via CBCT
  Other Names: Bio C-Temp
  Arms: Metapaste Calcium Hydroxide
Other: Bio C-Temp — Bio C-Temp
  Arms: Bio C-Temp

SUMMARY:
Periapical lesions are the commonly occurring pathologic lesions that affect the periradicular tissues of the tooth.This lesion can be classified as granuloma, cystic, or abscess .The pathological changes seen in some periradicular and periapical cases are due to the presence of microorganisms, and their byproducts.These released toxins have the ability to diffuse through inflamed pulpal tissue and get into the periapical area. In a necrotic pulp, the lack of blood flow in the root prevents host immunity from eliminating the infection.

DETAILED DESCRIPTION:
Endodontic treatment is essentially directed towards the prevention and control of pulpal and periradicular infections. Complete chemomechanical preparation may be considered an essential step in root canal disinfection. However total elimination of bacteria is difficult to accomplish. by remaining in the root canal between appointments, intracanal medicament may help to eliminate bacteria.

A medicament is an antimicrobial agent that is placed inside the root canal between treatment appointments in an attempt to destroy remaining microorganisms and prevent reinfection Thus, they may be utilized to kill bacteria, reduce inflammation (and thereby reduce pain), help eliminate apical exudate, control inflammatory root resorption and prevent contamination between appointments.When intracanal medicaments were not used between appointments, bacterial numbers increased rapidly.

The BIO-C® TEM has emerged as the first intracanal bioceramic medication of Endodontics, indicated for cases of treatment and retreatment due to its high pH to its antibacterial, bacteriostatic, anti- inflammatory and mineralization- -inducing action. Since it is a bioactive product, BIO-C® TEMP interacts with the surrounding tissue, stimulating healing. The tissue system responds to the material as if it was a natural tissue.

It has found its way in treatment of diverse cases: pulpitis, pulp necrosis, periapical lesion, persistent fistula, inflammatory or purulent exudate, perforation, apexification, external and internal resorption. It has been recommended not only for its actions, but also because it is a ready-to-use syringe, easy to insert into the root canal and with no painful symptomatology, even in cases where it has been extruded through the apical foramen.

Gradual release of Ca2+ Periodic exchange is not required, Biocompatible( Absence of symptomatology), High alkalinity (pH ~12)( Unsuitable environment for bacterial growth), Easy to remove( Clinical time optimization),and High radiopacity (Excellent radiographic visualization).

The intra-canal procedures based on the maximum elimination of the irritant including antimicrobial intra-canal dressing are valuable tool to control endodontic infections and theoretically prevent postoperative pain.

Periapical lesions, inflammatory reactions caused by bacterial infections in the periapical area of teeth, require effective treatment for optimal healing.For decades non-setting Ca(OH)2 has been the gold standard intracanal medicament in endodontic procedures to promote the healing of periapical lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mature teeth.
* Patients with periapical periodontitis.
* Maxillary anterior teeth only will be involved.
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
* Patients who will agree to the consent and will commit to follow-up period

Exclusion Criteria:

* Patients with immature roots.
* Patients with any systemic disease that may affect normal healing.
* Patients with swelling.
* Pregnant females.
* Patients who could/would not participate in a 1-year follow-up.
* Patients with old age.
* Teeth with periodontal involvement.
* Teeth with vertical root fractures.
* Non-restorable teeth.
* Cases with previously initiated endodontic treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Treatment of Postoperative Pain | from 0 hours to 2 weeks after the procedure
  Patients will be evaluated for postoperative pain via (NRS) to record the intensity of pain.as follows: 0 reading represents "no pain" ; 1- 3 reading represents "mild pain" ; 4- 6 reading represents "moderate pain" and 7- 10 reading represents "severe pain".

SECONDARY OUTCOMES:
Periapical Healing | After 6 months to 12 months
  Periapical healing will be evaluated by comparing the size of the initial lesion pre-operatively and postoperatively (after 6 and 12 months), using periapical radiographs and CBCT. This will be aggregated in percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Wael HUESSIEN KAMEL, Professor, Study Chair — Department of Endodontics, Faculty of Dentistry,Al-Azhar University
Locations (1):
- Minia University, Faculty of Dentistry, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No